CLINICAL TRIAL: NCT02775461
Title: Pancreas Disease and High Risk Registry
Brief Title: Pancreas Registry and High Risk Registry
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Aimee Lucas, Associate Professor, Gastroenterology, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 13-0222
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pancreas Cancer; Pancreatitis; Chronic Pancreatitis; Pancreatic Cyst; Family History of Pancreas Cancer; Genetic Mutations
Keywords: Pancreas Cancer; Chronic Pancreatitis; Pancreatic Cyst; BRCA1; BRCA2; Lynch Syndrome; Peutz-Jeghers syndrome; ATM mutation; FAMMM Syndrome; Pancreatitis; Family History of Pancreas Cancer; Family History of Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Pancreatitis, Chronic; Pancreatic Cyst; Colorectal Neoplasms, Hereditary Nonpolyposis; Peutz-Jeghers Syndrome; Melanoma, Cutaneous Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole Blood samples for DNA, serum and plasma extraction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hereditary Pancreas Cancer Syndrome: Patients that have a diagnosis or any family history of a hereditary pancreas cancer syndrome, such as, but not limited to, Familial Pancreatic Cancer, hereditary pancreatitis, FAMMM syndrome, FAP and its variants, HNPCC (Lynch syndrome), Peutz-Jeghers syndrome, or BRCA1 and/or BRCA2 germline mutations.
- Personal or FHx of Pancreas Cancer or Pancreas Cysts: Patients that have personal or family history of pancreatic cancer or pancreatic cysts.
- Inflammatory Pancreatic Diseases: Patients that have a personal or family history of pancreatic dysplasia or inflammatory pancreatic diseases.

SUMMARY:
The purpose of this study is to establish a registry of patients with pancreatic diseases. Patients included in the registry may include those with: pancreatic cancer, precancerous lesions of the pancreas, inflammatory lesions of the pancreas, cystic lesions of the pancreas, and patients at high-risk of pancreatic cancer such as those with a family history of pancreatic cancer or with a family history of a syndrome known to be associated with pancreatic cancer. Pancreatic cancer is the fourth leading cause of death from cancer in the United States. However, little is known about the development of pancreatic cancer and pancreatic diseases in individuals with the above conditions. Knowledge of how family history, environmental exposures, and inflammatory lesion of the pancreas contribute to the development of pancreatic cancer and pancreatic diseases is essential.

You may qualify to take part in this research study because you have inflammation in the pancreas, a pancreatic cyst, pre-cancerous lesions of the pancreas, pancreatic cancer, a family history of pancreatic cancer, or a family history of a syndrome known to be associated with pancreatic cancer.

We will also be collecting a blood sample from all participants for DNA isolation. Sometimes we are born with genes or DNA that give us an increased or decreased chance of developing an illness later in life. Genetic material will be isolated from your blood for further study. You may also choose to provide additional blood samples for serum and plasma extraction. Serum and plasma are components of the blood which can be used to measure indicators of disease in the blood, called biomarkers,for pancreatic diseases. Clinical data and biological specimens contained in this study may be used for a wide variety of future related studies to the cause, diagnosis, outcome and treatment of pancreatic cancer.

Funds for conducting this research are provided by Mount Sinai.

DETAILED DESCRIPTION:
The overall purpose of this research project is to establish a registry of patients with pancreatic diseases. Patients included in the registry may include those with: pancreatic cancer, precancerous lesions of the pancreas such as intraductal papillary mucinous neoplasms (IPMNs) and cystic lesions, inflammatory lesions and inflammation of the pancreas, and patients at high-risk of pancreatic cancer such as those with a family history of pancreatic cancer or with a family history of a syndrome known to be associated with pancreatic cancer. The data contained in this registry will be used to conduct research related to the risk of pancreatic cancer and pancreatic diseases. As this is a registry protocol, no specific hypotheses are to be tested.

Specific Aims:

1. Establish and maintain a registry of individuals and their family members who have pancreatic diseases and may be at increased risk of developing pancreatic cancer over normal population risk.
2. Collect data and review existing data on personal and family histories, demographics, risk factors, and health behaviors.
3. Use the data in the registry to conduct studies related to disease risk, prevention, and prognosis of pancreatic cancer and other pancreatic diseases.

Pancreatic cancer is the fourth leading cause of death from malignancy in the United States. With near equivalent incidence and mortality, cure can only be achieved with surgical resection of an early stage lesion. Premalignant disease stages, such as IPMN, may be detected with noninvasive and minimally invasive techniques, providing an opportunity for screening and surveillance of at-risk populations.

Knowledge of the etiology of pancreatic cancer is incomplete. Approximately 10% of pancreatic ductal adenocarcinoma (PDAC) has a hereditary component, and screening this population has the potential to have an impact on disease mortality. Certain patient populations, such as those with hereditary pancreatitis, Peutz-Jeghers syndrome, familial atypical multiple mole melanoma (FAMMM syndrome), Lynch syndrome, and the breast ovarian cancer syndrome (BRCA1 and BRCA2 mutations) are at the highest risk of PDAC. BRCA2 mutations are the most commonly identified germline mutations in families with PDAC. Even a family history of PDAC without the above described syndromes has been shown to increase risk, suggesting a unique familial pancreatic cancer syndrome which may be related to the partner and localizer of BRCA2 (PALB2) gene or other PDAC susceptibility genes. Environmental risk factors, such as cigarette smoking, diabetes, obesity and dietary risk factors have been implicated in the development of PDAC.

A sequential model of acquisition of somatic mutations via a Pancreatic Intraepithelial Neoplasia (PanIN) has been proposed for the development of PDAC and subsequent metastases. However, others have proposed that the metastatic process may be initiated earlier in the disease process during the pre-malignant cyst or PanIN phase. This may in part account for the fact that the overwhelming majority of patients diagnosed with PDAC are diagnosed when the lesion is already metastatic.

Several groups have instituted PDAC screening for individuals at high-risk of PDAC. These groups have demonstrated the feasibility of detection of PDAC and pre-malignant lesions in certain high-risk individuals. Given the large gaps in knowledge, recruitment of patients with preneoplastic pancreatic diseases to registries is essential in the development of effective PDAC screening and prevention programs.

As an increasing number of patients undergo cross-sectional imaging with the abdomen with cat scan (CT) and magnetic resonance imaging (MRI), an increasing number of patients are found to have pancreatic disease and pancreatic cysts. While there is an increased risk of pancreatic cancer with these lesions, the studies to date are small and retrospective.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 first degree relative affected with Pancreatic Cancer
* Any of (BRCA1, BRCA2, PALB2, ATM) mutations + 1 family member with Pancreatic Cancer
* mFAMMM (p16,CDKN2A mutations) + 1 family member with Pancreatic cancer
* Known mutation carrier for STK11 (Peutz Jeghers Syndrome)
* Lynch syndrome (HNPCC) + 1 family PDAC
* Known mutation carrier for Hereditary pancreatitis
* Individuals with a history of pancreatic cyst(s) (IPMN's) that measure ≥ 1 cm

Exclusion Criteria:

* Patients who do not speak English or Spanish
* Refusal by patient
* Individuals under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with inflammation in the pancreas, a pancreatic cyst, pre-cancerous lesions of the pancreas, pancreatic cancer, a family history of pancreatic cancer, or a family history of a syndrome known to be associated with pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1368 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Number of individuals with pancreatic diseases | 10 years
  Number of individuals and their family members who have pancreatic diseases and may be at increased risk of developing pancreatic cancer over normal population risk.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Lucas, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York